CLINICAL TRIAL: NCT02501083
Title: Natural History of Cardiac and Respiratory Function in Patients With Muscular Dystrophies on Home Mechanical Ventilation
Brief Title: Natural History of Cardiac and Respiration Function in Patients With Muscular Dystrophies on Home Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: CRHF-MD
Record Dates: First submitted 2015-06-26; First posted 2015-07-17 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Heart, Respiratory, Disease, Functional
Keywords: cardiomyopathy; echocardiography; prognosis; respiratory; home mechanical ventilation; vital capacity; maximal inspiratory pressure; maximal expiratory pressure
MeSH Terms: conditions — Disease; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — The study will not include any intervention.

SUMMARY:
Muscular dystrophies are inherited disorders that affect skeletal muscle. Cardiac and respiratory function may be affected in this group of diseases. The investigators sought to analyze the long term cardiac and respiratory function in patients with muscular dystrophies recquiring home mechnaical ventilation .

DETAILED DESCRIPTION:
Muscular dystrophies are neuromuscular disorders with disability and can affect respiratory muscle function and left ventricular function. Medical management of patients with cardiomyopathy relies mainly on angiotensin-converting-enzyme inhibitors and beta blockers. Respiratory management relies on home mechanical ventilation and couph assist.

The investigators aim

* to analyze cardiac and respiratory function over time in patients with muscular dystrophies followed at the home mechanical ventilation unit.
* to determine the long term impact of the home mechanical ventilation on cardiac and respiratory events and to define the predictive factors associated.

Patients will be included retrospectively. Tissue Doppler imaging and Tricuspid annular plane systolic excursion were used for the assessment of the right ventricle. Left ventricular ejection fraction was used for the analysis of the left ventricle. Respiratory function was assessed using the vital capacity, the maximal inspiratory pressure, the maximal expiratory pressure, the peak couph flow rate.

ELIGIBILITY:
Inclusion Criteria:

* Age higher or equal to 18 years
* Duchenne muscular dystrophy
* Becker muscular dystrophy
* Sarcoglycanopathy
* limb girdle muscular dystrophy
* Pompe disease
* Steinert disease
* FSH disease
* Others myopathies

Exclusion Criteria:

* Minor patient
* Sepsis condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with muscular dystrophies
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
predictive factors for long term survival | 10 years

SECONDARY OUTCOMES:
predictuve factors for cardiac events | 10 years
predictive factors for respiratory events | 10 years
cumulative cardiac events incidence | 10 years
cumulative respiratory events incidence | 10 years
annual rate of left ventricular ejection fraction decline | 10 years
annual rate of respiratory vital capacity decline | 10 years
annual rate of maximal inspiratory pressure decline | 10 years
annual rate of maximal expiratory pressure decline | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah FAYSSOIL, MDPhD, Principal Investigator — HOPITAL RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, France

REFERENCES:
- [Derived] Fayssoil A, Mansencal N, Nguyen LS, Nardi O, Yaou RB, Leturcq F, Amthor H, Wahbi K, Becane HM, Lofaso F, Prigent H, Bassez G, Behin A, Stojkovic T, Fontaine B, Duboc D, Dubourg O, Clair B, Laforet P, Annane D, Orlikowski D. Prognosis of Right Ventricular Systolic Dysfunction in Patients With Duchenne Muscular Dystrophy. J Am Heart Assoc. 2023 Aug 15;12(16):e027231. doi: 10.1161/JAHA.122.027231. Epub 2023 Aug 10. PMID 37581390
- [Derived] Fayssoil A, Lazarus A, Wahbi K, Ogna A, Nardi O, Lofaso F, Clair B, Orlikowski D, Annane D. Cardiac implantable electronic devices in tracheotomized muscular dystrophy patients: Safety and risks. Int J Cardiol. 2016 Nov 1;222:975-977. doi: 10.1016/j.ijcard.2016.08.040. Epub 2016 Aug 6. PMID 27526372
- [Derived] Fayssoil A, Ogna A, Chaffaut C, Chevret S, Guimaraes-Costa R, Leturcq F, Wahbi K, Prigent H, Lofaso F, Nardi O, Clair B, Behin A, Stojkovic T, Laforet P, Orlikowski D, Annane D. Natural History of Cardiac and Respiratory Involvement, Prognosis and Predictive Factors for Long-Term Survival in Adult Patients with Limb Girdle Muscular Dystrophies Type 2C and 2D. PLoS One. 2016 Apr 27;11(4):e0153095. doi: 10.1371/journal.pone.0153095. eCollection 2016. PMID 27120200